CLINICAL TRIAL: NCT05694988
Title: An Open Controlled Randomized Study of the Efficacy and Safety of the Method of Combined Use of Non-selective Hemosorption (Efferon CT) and High Volume Hemofiltration (HVHF) in Patients With Acute Pancreatitis.
Brief Title: Combination of Cytokine Hemosorption and High-volume Hemofiltration in Acute Pancreatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-ct-2022-03
Record Dates: First submitted 2023-01-13; First posted 2023-01-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Pancreatitis Without Necrosis or Infection
Keywords: acute pancreatitis; sepsis; cytokines apsorbtion; hemoperfusion
MeSH Terms: conditions — Infections; Pancreatitis; Sepsis

STUDY DESIGN:
Intervention Model Description: The study will be randomized stratified 1:1. The stratification criterion is the patient's SOFA index score.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline therapy (No Intervention): Basic therapy - the routine practice of an institution for the treatment of patients with uninfected acute pancreatitis
- Basic therapy + Efferon CT + HVHF (Experimental): Basic therapy, which is the routine practice of an institution for the treatment of patients with acute nonseptic pancreatitis in combination with extracorporeal hemoperfusion therapy (Efferon CT) and high-volume hemofiltration (HVHF).
  Interventions: Device: Efferon CT

INTERVENTIONS:
Device: Efferon CT — Efferon CT (JSC Efferon, Moscow, RF) is a device for extracorporeal blood purification by direct hemoperfusion. Detoxification is carried out by sorption of cytokines and other products of endogenous intoxication with a molecular size of up to 55 kDa.
  Arms: Basic therapy + Efferon CT + HVHF

SUMMARY:
Mortality from severe acute pancreatitis reaches 42%. The prognosis of acute pancreatitis is associated with the development of acute inflammatory response syndrome (SIRS) and multiple organ failure (MOF). Due to the lack of etiological therapy, the treatment of acute pancreatitis is predominantly symptomatic.

Severity and mortality are associated with early systemic inflammatory response syndrome (SIRS) and septic complications in the later stages of the disease.

In connection with a pronounced inflammatory reaction ("cytokine storm") in the early phase of endogenous intoxication of acute pancreatitis, a promising therapeutic approach is the extracorporeal removal of cytokines.

This prospective study intends to study the effect of hemoperfusion (Efferon CT) in combination with high-volume hemofiltration (HVHF) on the severity of symptoms of endogenous intoxication and indicators of organ dysfunction in acute pancreatitis.

DETAILED DESCRIPTION:
Acute pancreatitis in emergency surgery ranks third in frequency of its manifestation, second only to acute appendicitis and cholecystitis. The incidence of acute pancreatitis is growing from year to year and is more than 38 patients per 10,000 population per year. In 25% of patients, the development of pancreatitis is destructive.

Mortality in this pathology is mainly associated with the development of severe necrotic forms that cause a systemic inflammatory response of the body. The formation of pancreatic necrosis occurs within 1-2 days of illness, and it is at this time that the therapeutic effect is most effective.

Mortality in patients with acute pancreatitis reaches 20-60% depending on the nature of the disease, the phase of the pathological process, the severity of concomitant diseases, the severity of multiple organ failure syndrome (MODS), purulent-septic complications, and the development of septic shock. The main factors determining an unfavorable prognosis are the frequency of multiple organ failure and the development of sepsis, their intensity, as well as the developed septic shock. In the case of the onset and progression of multiple organ failure in the first 48 hours, they speak of early severe pancreatitis, which is characterized by a more unfavorable prognosis.

Acute pancreatitis is a systemic rather than a local critical condition. Associated complications include sepsis, multiple organ failure, ARDS, acute renal failure, disseminated intravascular coagulation syndrome, acute liver failure, etc. According to some reports, at least 50% of deaths in the early stage of acute pancreatitis are associated with multiple organ failure, and failure of three or more organs, mortality rises to 95%.

The moment when timely treatment can affect the outcome of the disease is often missed. Against the background of a picture of developed pancreatic necrosis, complications arise at lightning speed, despite the measures taken to prevent them.

The earliest possible detection of patients with an aggressive, destructive nature of the disease is very important for the entire complex of intensive care. The severity of the patient's condition with acute pancreatitis is largely determined by the severity of endotoxemia. The latter, in turn, depends on the cytokine response of the body.

To date, the early pathogenetic mechanisms of acute pancreatitis and its complications have not been sufficiently studied. The question of what happens at the subcellular level, what processes are responsible for the development of severe forms of the disease, extraorganic complications, remains insufficiently studied.

Treatment of acute pancreatitis is traditionally divided into conservative and surgical. The start time of conservative measures, their components, an adequate assessment of effectiveness affect the timing and extent of surgical intervention.

At the moment, there is no specific surgical approach for sterile and infected pancreatic necrosis. It is known that mortality from infected pancreatic necrosis is 2-3 times higher than from a sterile process.

"Cytokine storm", which occurs in the acute phase of pancreatitis, leads to aggravation of intoxication, inadequate and untimely correction of which underlies the development of pancreatogenic shock, multiple organ failure and septic complications.

Organ hypoperfusion, tissue hypoxia, endotoxicosis, systemic inflammatory and anti-inflammatory reactions induced by "mediator aggression" and electrolyte disturbances are the most important links in the etiopathogenesis of acute pancreatitis and multiple organ failure. Therefore, the use of detoxification methods aimed at removing toxic substances, normalizing organ perfusion, reducing systemic inflammation in the treatment of patients with acute pancreatitis is pathogenetically justified in order to prevent multiple organ failure, pancreatic shock and sepsis.

In the last 10 years, various methods of extracorporeal detoxification have become widespread in the practice of intensive care for severe forms of acute pancreatitis.

Nevertheless, there is no consensus among specialists regarding the timing of the application of certain methods, taking into account the phase course of acute pancreatitis, the required frequency of procedures and their effectiveness.

In acute pancreatitis, severe endotoxemia occurs early, leading to multiple organ failure. Allocate biochemical, immunological and microbial components of endogenous intoxication, which include intermediate and final metabolites of the processes of autolysis and secondary infection.

Detoxification underlies the prevention and pathogenetic treatment of complications of acute pancreatitis. Numerous studies have shown that the use of extracorporeal sorption methods that eliminate pro-inflammatory cytokines improves the results of treatment of patients with manifestations of endogenous intoxication.

Accumulated evidence in recent years suggests that continuous veno-venous hemofiltration is beneficial in acute pancreatitis by removing inflammatory molecules and medium and low molecular weight toxic substances by convection. Particular attention is paid to high-volume hemofiltration, which can give a better effect in the treatment of acute pancreatitis.

The 2012 study by La-Ping Chu (China) "Clinical effects of pulsed high-volume hemofiltration in severe acute pancreatitis complicated by multiple organ dysfunction syndrome" also confirmed that high-volume hemofiltration has a pronounced beneficial effect on clinical symptoms and laboratory parameters in acute pancreatitis with multiple organ failure .

In acute pancreatitis, a large number of soluble inflammatory mediators circulate in the patient's blood. Thus, the elimination of cytotoxins with standard continuous hemofiltration with a water exchange rate of 35 ml/kg/h may not be adequate for the severity of symptoms of the disease. The advantage of "high volume" is the removal of substances with a higher molecular weight, which include many inflammatory mediators. Numerous animal studies have shown a positive effect of high volume hemofiltration (HVHF) on survival in endotoxic models. Human studies have shown that HVHF improves hemodynamics in septic shock. But the great concern of researchers has always been the difficulty of performing high-volume hemofiltration as a continuous method. That is why it is of interest to study the effectiveness of short-pulse hemofiltration techniques in acute pancreatitis.

Recently, a search is underway for new approaches to the treatment of patients in the early stages of acute pancreatitis, even before the development of severe complications that significantly worsen the prognosis of the disease. One of them may be the extracorporeal removal of excessively produced inflammatory mediators (cytotoxins) from the systemic circulation by sorption. Nevertheless, very few studies have been devoted to the use of the hemosorption method in the early stage of acute pancreatitis, before the appearance of purulent-septic complications.

Hemosorption is a modern method of removing from the patient's blood substances that are toxic to body cells. Currently, there are no multicenter randomized studies confirming the need to use extracorporeal therapy methods as one of the main areas of pathogenetic therapy for acute pancreatitis. At the same time, there is more and more evidence of a significant effect of an increase in the level of cytokines on the pathogenesis of the disease and its progressive deterioration, which suggests a possible positive role of the cytokine hemosorption method performed in the early phase of acute pancreatitis.

In connection with the above data, it seems interesting to determine the degree of influence of the combined method of cytokine hemosorption (Efferon CT) and high-volume hemofiltration on the clinical manifestations of endogenous intoxication and organ dysfunction in acute pancreatitis. proceeding without septic complications.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years old,
* Acute pancreatitis according to the Atlanta classification of OP (2012), without signs of infection,
* Acute pancreatitis confirmed by tomography. Score according to the Modified CTSI Pancreatitis Severity Index: from 4 points and above,
* No more than 3 days from the onset of an attack of acute pancreatitis,
* APACHE II score - at least 10,
* The patient must receive adequate fluid therapy (at least 30 ml/kg) from the time of randomization until the first therapy,
* The patient's condition allows therapy for at least 4 hours.

Exclusion Criteria:

* Age over 75,
* More than 3 days from the onset of an attack of acute pancreatitis,
* An attack of acute pancreatitis, as an exacerbation of chronic pancreatitis.
* Acute pancreatitis as a complication of a surgical operation,
* DS - Septic shock (Sepsis-3, 2016)
* The presence of a focus of non-sanitized surgical infection,
* Charlson comorbidity index> 5 points,
* Critical hypoxemia (PaO2/FiO2 < 150 mm Hg),
* GCS level of consciousness < 12 points,
* Obesity 3 degrees and above (weight over 150 kg),
* Blood triglyceride level >1000 mg/dl, (11.2 mmol/l),
* Dementia,
* Inability to achieve or maintain min SBP ≥ 65 mm Hg. Art., despite vasopressor therapy and infusion therapy in tech. 24 hours
* Presence of end-stage renal disease requiring RRT,
* The presence of cirrhosis of the liver (> 5 points according to the Child-Pugh classification),
* Unresolved biliary hypertension syndrome,
* Acute thromboembolism of the pulmonary artery, confirmed by tomography,
* Acute myocardial infarction within the last 4 weeks,
* Acute cerebrovascular accident,
* Transfusion reaction,
* Severe congestive heart failure,
* Uncontrolled bleeding (acute blood loss in the last 24 hours).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect of the combined use of the Efferon CT device and HVHF on indicators of organ dysfunction | 1-72 hours
  The value of indicators on the SOFA scale every 24 hours ± 1 hour from the start of hemoperfusion (0 hour) to 72 hours.

SECONDARY OUTCOMES:
Effect of using the combined use of the Efferon CT device and HVHF on systemic hemodynamic parameters | 1-72 hours
  Time (number of hours) from randomization to end of vasopressor support.
Effect of the combined use of the Efferon CT device and HVHF on pulmonary oxygen metabolism function | 1-72 hours
  Value of oxygenation index (Pa02 / Fi02 (Pa) every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 72 hours.
Effect of the combined use of the Efferon CT device and HVHF on the indicators of the cardiac index | 1-72 hours
  Ultrasound assessment of LVOT VTI or RVOT VTI gain

CONTACTS AND LOCATIONS:
Overall Officials: Makariy Mendibaev, MD, Principal Investigator — Demikhov City Clinical Hospital of the Moscow Health Department
Locations (1):
- V.P. Demikhov City Clinical Hospital No. 68, Moscow, Russia